CLINICAL TRIAL: NCT02920671
Title: Skeletal Muscle Oxidative Phosphorylation Capacity and Nutrient Homeostasis in Individuals With Primary (Genetic) and Secondary (Obesity-related) Mitochondrial Impairment as Compared to Healthy, Normal-weight Individuals
Brief Title: Muscle OXPHOS and Nutrient Homeostasis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 825558
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Mitochondrial Diseases; Obesity
MeSH Terms: conditions — Mitochondrial Diseases; Obesity | interventions — Glucose Tolerance Test; Absorptiometry, Photon; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood will be collected as part of this protocol. Results from screening laboratory studies will be entered into the secure database, and copies will be sent to the participant, as well as his/her physician if s/he wishes.
  De-identified, specimens coded with the participant's ID number will be stored in anticipation of future studies.
  DNA/RNA will be extracted and stored pending future analyses to be specified (e.g., whole exome or mitochondrial DNA sequencing, gene expression studies). No results of genetic analyses will be included in the electronic medical record. Participants will not be informed of results.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mitochondrial Disease: Clinical history consistent with the diagnosis of mitochondrial disease, and molecular genetic diagnosis.
  Interventions: Other: Tracer-enhanced oral glucose tolerance test (OGTT*); Other: Muscle MRI; Other: Dual energy x-ray absorptiometry (DXA); Other: Questionnaires
- Obese: BMI > 30 kg/m2. These will be matched with subjects with mitochondrial disease by age, sex, estrogen status (women), and usual self-reported physical activity.
  Interventions: Other: Tracer-enhanced oral glucose tolerance test (OGTT*); Other: Muscle MRI; Other: Dual energy x-ray absorptiometry (DXA); Other: Questionnaires
- Normal Weight & Overweight: BMI 18.5 - < 30 kg/m2. These will be matched with subjects with mitochondrial disease by age, sex, estrogen status (women), and usual self-reported physical activity.
  Interventions: Other: Tracer-enhanced oral glucose tolerance test (OGTT*); Other: Muscle MRI; Other: Dual energy x-ray absorptiometry (DXA); Other: Questionnaires

INTERVENTIONS:
Other: Tracer-enhanced oral glucose tolerance test (OGTT*) — Oral glucose tolerance test with stable isotope tracers will be administered. Resting energy expenditure and respiratory quotient will be evaluated during this test using indirect calorimetry.
Other: Muscle MRI — Non-invasive muscle MRI will be performed to evaluated metabolic capacity.
Other: Dual energy x-ray absorptiometry (DXA) — DXA will be performed to evaluate body composition.
Other: Questionnaires — Questionnaires will be used to evaluate participants' health and habits.

SUMMARY:
Investigators are recruiting adults (men and women, ages 18 to 65 years, inclusive) with a confirmed genetic diagnosis of mitochondrial disease. Investigators are also recruiting both obese and normal-weight healthy volunteers (men and women, ages 18 to 65 years, inclusive) without a family history of mitochondrial disease to compare to affected individuals.

The study involves non-invasive MRI methods and glucose tests to focus on the relationship between mitochondrial disease, obesity, and the risk of diabetes. All study visit procedures will be completed within 2 days, which includes an overnight stay at the Hospital of the University of Pennsylvania. There are no study medications or sedations, and participants will be continually monitored during minimally-invasive procedures (e.g., blood draws).

All participants will be able to receive compensation. Furthermore, it may be possible to provide reimbursement for travel, lodging, and meals for individuals with mitochondrial disease.

Investigators hope that this research will contribute to the current knowledge of mitochondrial disease and that it will improve diagnostic and treatment approaches.

DETAILED DESCRIPTION:
Although obesity is a significant public health problem, why obesity leads to diabetes in some individuals but not others is poorly understood. Mitochondrial impairment, particularly in skeletal muscle with its high energy requirement, has been implicated in the pathogenesis of obesity-related insulin resistance. In addition, individuals with genetic disorders affecting mitochondrial function are at increased risk of diabetes. The proposed studies will investigate the association between skeletal muscle oxidative phosphorylation capacity (OXPHOS), which is a dimension of mitochondrial function, and glucose and lipid homeostasis in (i) individuals with genetic disorders of muscle mitochondrial function as compared to (ii) non-obese adults and (iii) otherwise healthy obese adults.

During a single 2-day, 1-night study visit, investigators will use innovative, non-invasive magnetic resonance imaging-based methods of estimating skeletal muscle oxidative phosphorylation capacity, including post-exercise chemical exchange saturation transfer (CrCEST) recovery and 31-Phosphorus (31P) magnetic resonance spectroscopy (MRS) and muscle lipid content, including 1H magnetic resonance spectroscopy (MRS) and 3-point Dixon techniques, in conjunction with a tracer-enhanced oral glucose tolerance test (OGTT*) to measure overall insulin sensitivity and the selective effect of insulin on glucose disposal (Rd). The percentage suppression of endogenous glucose production by the oral glucose load (% suppression of Ra of endogenous glucose) will also be assessed. Infusion of a glycerol tracer permits assessment of lipolysis in both the fasting state, and also after the oral glucose load, such that the percentage suppression of lipolysis by the oral glucose load can also be calculated (% suppression of Ra of glycerol). In addition, the insulin and c-peptide minimal models will also be used to model pancreatic β-cell responsiveness to the oral glucose load and hepatic insulin extraction.

ELIGIBILITY:
Inclusion Criteria:

Indvidiuals who meet all of the following criteria are eligible for participation in the study:

1. Male and female patients age 18 to 65 years of age.
2. Ability to provide written informed consent.
3. Cognitively and medically stable and able to comply with the procedures of the study protocol.

For individuals with mitochondrial disease:

Clinical history consistent with the diagnosis of mitochondrial disease, and molecular genetic diagnosis. To ensure consistency with other trials performed in mitochondrial disease, investigators will also ensure that participants meet the same set of previously published criteria. These include clinical features consistent with primary mitochondrial disease and molecular genetic proof of a pathogenic mutation in mtDNA or nDNA in a gene known to be associated with dysfunction of complexes I-V of the respiratory chain. Specifically, eligible participants must have defined mtDNA or nDNA mutations affecting subunits or assembly of these complexes that are associated with known clinical/pathological features, such as chronic progressive external ophthalmoplegia (CPEO), Kearns-Sayre, mitochondrial encephalomyopathy, lactic acidosis and stroke-like episodes (MELAS), mitochondrial encephalopathy and ragged red fibers (MERRF), neuropathy, ataxia and retinitis pigmentosa (NARP) or Leigh syndrome (45). Investigators will explicitly include individuals with Friedreich's Ataxia (46), a mutation in the mitochondrial protein frataxin, and those with mutations in respiratory chain complex II protein, succinate dehydrogenase (SDH).

For normal weight participants:

BMI < 25 kg/m2. These will be matched with subjects with mitochondrial disease by age, sex, estrogen status (women), and usual self-reported physical activity (as either sedentary or not, i.e., for sedentary, less than 30 minutes of moderate physical activity 5 days per week, or vigorous physical activity for 20 minutes 3 days per week).

For obese participants:

BMI > 30 kg/m2. These will be matched with subjects with mitochondrial disease by age, sex, estrogen status (women), and usual self-reported physical activity (as either sedentary or not, i.e., for sedentary, less than 30 minutes of moderate physical activity 5 days per week, or vigorous physical activity for 20 minutes 3 days per week).

Exclusion Criteria:

For all study groups (i.e., mitochondrial disease, normal weight, obese):

1. Diabetes (HgbA1c > 6.4%) and/or taking insulin or other anti-diabetic drug therapy within the 4 weeks prior to enrollment.
2. Use of any lipid-lowering medication (excluding nutritional supplements) within the 4 weeks prior to enrollment.
3. Any contraindication to MRI study (e.g., implanted non-compatible device, pacemaker, known claustrophobia).
4. Kidney disease. Estimated glomerular filtration rate < 60 ml/min/1.73 m2 (calculated using the subject's measure serum creatinine and the Modification of Diet in Renal Disease [MDRD] study estimation formula).
5. Liver disease. Persistent elevation of liver function tests at the time of study entry. Persistent SGOT (AST), SGPT (ALT), Alk Phos or total bilirubin, with values > 3 times normal upper limits, will exclude a subject from study participation.
6. Severe co-existing cardiac disease, characterized by any one of these self-reported conditions:

   1. recent myocardial infarction (within the past 6 months).
   2. evidence of ischemia on functional cardiac exam within the last year
   3. left ventricular ejection fraction < 30%.
7. Acute or chronic pancreatitis.
8. Receiving treatment for a medical condition requiring chronic use of systemic (oral or parenteral steroids, except for the use of < 5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
9. Anemia (baseline hemoglobin concentration < 11 g/dl in women and <12 g/dl in men), lymphopenia, (< 1,000/µL), neutropenia (< 1,500/µL), or thrombocytopenia (platelets < 100,000/µL).
10. Any known coagulopathy (including Factor V deficiency) or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) (low-dose aspirin treatment is allowed) or patients with an INR > 1.5.
11. For female participants: Positive pregnancy test.
12. Known active alcohol or substance abuse, including known tobacco use.
13. Use of any investigational agents within 4 weeks of enrollment.
14. Inability to fast comfortably for 10 hours (i.e., overnight).
15. Individuals who have a pacemaker, metal implants, claustrophobia, have worked around a metal grinder or a construction site, or that have known medical conditions which can be exacerbated by stress such as anxiety or panic attacks. Inability to lie flat in the MRI scanner for 90 minutes is also an exclusion criterion.

    In addition, specific exclusion criteria for undergoing MRI scanning include:
    * ANY intra-luminal implant, filter, stent or valve replacement
    * ANY type of life assist device, pump, or prosthetic
    * ANY vascular clip or clamp
    * ANY surgically placed clips or clamps or bands on visceral organs
    * ANY intracranial implants of any type other than dental fillings
    * ANY non-removable piercings, jewelry, or medicinal patch
    * ANY personal history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic examination.
    * ANY personal history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation.
16. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll three groups of individuals (mitochondrial disease, obese, normal weight).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Glucose rate of disposal (glucose Rd) during OGTT* | 1 day
  The primary outcome for the present study will be glucose rate of disposal (Rd) during the OGTT*

SECONDARY OUTCOMES:
Exogenous rate of glucose appearance (exogenous glucose Ra) during OGTT* | 1 day
Endogenous rate of glucose appearance (endogenous glucose Ra) during OGTT* | 1 day
Endogenous rate of glycerol appearance (endogenous glycerol Ra) during OGTT* | 1 day
Post-exercise exponential time constant for decline in CrCEST (skeletal muscle MRI) | 1 day
Resting CrCEST (skeletal muscle MRI) | 1 day
Muscle fat content (skeletal muscle MRI) | 1 day
Blood glucose variability (continuous glucose monitoring) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Shana McCormack, MD, MTR, Principal Investigator — University of Pennsylvania & Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Tamaroff J, Nguyen S, Wilson NE, Stefanovski D, Xiao R, Scattergood T, Capiola C, Schur GM, Dunn J, Dedio A, Wade K, Shah H, Sharma R, Mootha VK, Kelly A, Lin KY, Lynch DR, Reddy R, Rickels MR, McCormack SE. Insulin Sensitivity and Insulin Secretion in Adults With Friedreich's Ataxia: The Role of Skeletal Muscle. J Clin Endocrinol Metab. 2025 Jan 21;110(2):317-333. doi: 10.1210/clinem/dgae545. PMID 39109797